CLINICAL TRIAL: NCT01633996
Title: Effectiveness of Acupuncture Augmentation on Treatment Resistant Depressed Patients
Brief Title: Effectiveness of Acupuncture for Depressed Patients Taking Antidepressant Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Albert Yeung, Director of Primary Care Research, Depression Clinical and Research Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002-P-001899
Record Dates: First submitted 2012-06-15; First posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Depression
Keywords: Acupuncture; Antidepressant; Augmentation; Depression
MeSH Terms: conditions — Depression | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acupuncture (Experimental): All participants received open acupuncture augmentation treatment per the uniform acupuncture treatment protocol that we developed according to Traditional Chinese Medicine (TCM) principles for treating depression (see Intervention Description).
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Our acupuncture treatment protocol included: HT-7 and LI-4 on the hands bilaterally, and ST-36, SP-6, and LR-3 on the legs bilaterally, with gentle manual tonification every 10 minutes; and GV-20 and GV- 24.5 (Yintang), along the midline of the head.

SUMMARY:
In this research study, the investigators piloted a uniform acupuncture treatment protocol among adults with depression who were taking an antidepressant medication that was providing only partial or no symptom alleviation. The study's aims were evaluate the efficacy, safety, and tolerability of acupuncture augmentation treatment among this population. The investigators hypothesized that acupuncture as an augmentation treatment would be associated with a response rate of at least 50%, which the investigators defined as a decrease in depressive symptoms from the beginning to the end of the study of 50% or more, and that the response would be greater among patients who received acupuncture 2 times per week (vs. 1 time per week). The investigators also hypothesized that acupuncture would be associated with minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* A HAM-D-17 score of >= 14
* Partial or nonresponse to a standard antidepressant (monotherapy or combination) at an adequate dose over the past 8 or more weeks (natural agents such as omega-3 fatty acids, St John's wort, SAMe, and folic acid, were allowed as antidepressants)
* Concurrent psychotherapy was allowed, provided that it was not initiated within the 3 months prior to study entry.

Exclusion Criteria:

* A primary diagnosis other than major depressive disorder, or any history of psychosis or mania
* Conditions that could make it difficult to conclusively determine that depressive symptoms were the result of major depression and not some other condition, including any form of substance abuse or dependence within the last 6 months, other medical conditions that could be the basis of a depression (including epilepsy, history of an abnormal EEG, severe head trauma, or stroke)
* Serious uncontrolled medical conditions (e.g. poorly controlled diabetes, severe congestive heart failure), or other medical conditions that had not been stable for at least 3 months
* Having had electroconvulsive therapy (ECT) during the past year
* Current active suicidal or self-injurious potential necessitating immediate treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Response to acupuncture augmentation treatment, defined as a change in scores on the Hamilton Depression Rating Scale, 17 items (HAM-D-17) from baseline to endpoint. | Baseline and all acupuncture sessions (weekly) for 8 weeks
  The HAM-D-17 is a clinician-rated measure of patient depressive symptoms (structured interview). Higher cumulative scores indicate more severe depression. A 50% or greater reduction in HAM-D-17 from baseline to endpoint was considered representative of our hypothesized acupuncture-augmentation response rate of at least 50%.

SECONDARY OUTCOMES:
Evidence of acupuncture augmentation's tolerability and acceptability, as determined clinically by the participant and study doctor. | Once per acupuncture session (weekly) for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yeung, MD, ScD, Principal Investigator — Depression Clinical and Research Program, Massachusetts General Hospital
Locations (1):
- Depression Clinical and Research Program, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Yeung AS, Ameral VE, Chuzi SE, Fava M, Mischoulon D. A pilot study of acupuncture augmentation therapy in antidepressant partial and non-responders with major depressive disorder. J Affect Disord. 2011 Apr;130(1-2):285-9. doi: 10.1016/j.jad.2010.07.025. Epub 2010 Aug 6. PMID 20692042